CLINICAL TRIAL: NCT02877901
Title: Effect of Long Acting Anticholinergic on Nocturnal Incontinence After Radical Cystectomy and Orthotopic Neobladder. A Randomized Placebo-controlled Crossover Study
Brief Title: Effect of Long Acting Anticholinergic on Nocturnal Incontinence After Radical Cystectomy and Orthotopic Neobladder
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mohamed Hassan Zahran, lecturer of urology, Mansoura University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Zahran MH17082016
Record Dates: First submitted 2016-08-17; First posted 2016-08-24 (Estimated); Last update posted 2017-12-27 (Actual); Status verified 2017-12

CONDITIONS: Nocturnal Incontinence

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- tolterodine-treated group (Active Comparator): they will receive long acting tolterodine 4 mg at bedtime for 4 weeks. After that re-evaluation. then stop medication for two weeks (washout period).
  Interventions: Drug: long acting tolterodine 4 mg
- placebo-control group (Placebo Comparator): they will receive placebo at bedtime for 4 weeks. After that re-evaluation. then stop for two weeks (washout period). Then re-evaluate the nocturnal incontinence status and crosed over to receive long acting tolterodine 4 mg for 4 weeks. at the end the nocturnal incontinence status will be evaluated
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: long acting tolterodine 4 mg — receive one tablet at bed time for 4 weeks
  Arms: tolterodine-treated group
Drug: placebo — one tablet at bed time
  Arms: placebo-control group

SUMMARY:
It is a prospective randomized- placebo control crossover study to evaluate the effect of long acting tolterodine (anticholinergic) in improving and treating nocturnal incontinence in patient after radical cystectomy and orthotopic urinary diversion. patients will be randomly allocated into two groups. one will receive the drug and the other will receive placebo. continence status will be evaluated before and 4 weeks after treatment by the number of pads used and the ICIQ-UI short form questionnaire. This is followed by two weeks of drug washout then reevaluation of the continence status and each group will be crossed over and lastly will be evaluated again.

DETAILED DESCRIPTION:
Introduction:

Radical cystectomy (RC) and urinary diversion remain the gold standard for treatment of muscle invasive bladder cancer.1 The optimal goal is to control the malignancy, preserve renal function and optimize health related quality of life. Decision of urinary diversion selection has been changed in the last three decades from non-continent diversion to orthotopic neobladder (ONB), to maintain voiding pattern closely similar to normal pattern and to improve the overall health related quality of life (HRQOL).2 However, the continence status after ONB is affected by many factors, such as patient's age, mental status, intact and innervated external urethral sphincter, the reservoir capacity and pressure, presence of infection and the completeness of voiding.3 The recovery of continence status takes from six to 12 months after the operation to achieve day time continence which is regained earlier than nocturnal continence which takes 12 to 24 months.3 The reported day time continence ranges from 85 to 90% and NI in most series ranges from 20 to 40%.4- 7 in women, the reported incidence of day time and NI ranged from 68 to 100% and 26 to 89%, respectively.8- 11 Nocturnal incontinence is a major problem that affect HRQOL . In a multicenter study, individuals with ONB and NI have lower HRQOL, 12 this is similar to our data on female patients with ONB.2 Nocturnal incontinence may be due to patient and pouch causes. Loss of afferent input from the Detrusor muscle to the central nervous system is thought to account for the worsening of nocturnal continence.13 In a study, done by El Bahnasawy et al, to evaluate the factors affecting the NI after RC and ONB; higher pressure, positive urine culture, large post voiding residual volume, decreased maximal urethral pressure, decreased flow rate and patient compliance are associated with higher incidence of NI. However, on multivariate analysis, only post voiding residual volumes, frequency, and maximal amplitude of uninhibited contractions remained significantly associated with NI.14 Fifty percent of women with NI after RC and ONB have had pouch hyperactivity on urodynamic evaluation.15 To optimize nocturnal continence, patients are recommended to avoid sleeping pills and alcohol in the evening, to void before going to sleep, and to set up an alarm to void at least once during the night. Also proper treatment of infection is recommended.3 Up to 25% of patients reported an improved nocturnal continence with the use of imipramine hydrochloride 25 mg at bedtime. 14,16In a prospective randomized crossover study comparing 20 male enuretic patients with ileal ONB receiving oxybutynin versus verapamil, both groups showed improved urodynamic parameters and nocturnal continence status in 70% and 55% of patients, respectively.17 Ali-El-Dein et al, reported that treatment of female patients, who have NI after RC and ONB, with anticholinergic drugs (tolterodine or oxybutynin chloride) has associated with improvement and cure of NI in 36% and 23%, respectively.15 These data confirmed the efficacy of the anticholinergic use in treatment of NI after RC and ONB.

In the current study, we will study the role of long acting anticholinergic (tolterodine 4 mg) at bedtime in management of NI after RC and ONB through a prospective randomized placebo-controlled crossover study.

Material and methods:

Patients:

All patients for whom RC and ONB and attend for routine follow up at the outpatient clinic of Urology and Nephrology Center will be evaluated for eligibility of inclusion in this study.

Study design:

A single center prospective randomized placebo-controlled crossover study. It will be held in Urology and Nephrology Center, Mansoura University after approval of the local ethical committee. Patients meet the inclusion criteria will be included in the study. All patients will be evaluated by proper history, examination, BMI, ICIQ-UI Short Form, urine culture, serum creatinine and abdominal and pelvic ultrasound. Patients with positive urine culture will be treated by the appropriate antibiotic treatment till urine became sterile. Then, patients will be randomly allocated in 2 groups (1:1) by computer generated random numbers. The first group will receive long acting tolterodine (Incont LA, Adwia, Egypt) 4 mg at bedtime. The second group will receive placebo at bedtime. Both groups will be maintained on medication for 4 weeks. After that, both groups will be exposed to a period of two weeks of washout then crossed over to the alternate therapy.

Patients will be assessed for nocturnal incontinence by the number of episodes per week, number of pad used and ICIQ-UI short form questionnaire at the beginning of the study, after 4 weeks, after washout period then at the end of the study.

The ICIQ-UI short form is developed for assessing the prevalence, severity, impact on quality of life, and type of UI.19 The three scored items of the ICIQ-UI SF are:

1. How often do you leak urine? (0 ''Never,'' 1 '' About once a week or less often,'' 2 ''Two or three times a week,'' 3 ''About once a day,'' 4 ''Several times a day,'' 5 ''All the time''),
2. How much urine do you usually leak (whether you wear protection or not)? (0 ''None ,'' 2 ''A small amount,'' 4 ''A moderate amount,'' and 6 ''A large amount'')
3. Overall, how much does leaking urine interfere with your everyday life? (Visual analogue scale ranging from 0 ''Not at all'' to 10 ''A great deal''). Additional question is used to determine when urine leakage occurs. The answers result in a sum, with minimum score of 0, and maximum score of 21. Preliminary cut-off scores were set to 0 = ''no incontinence'' and ˃1= ''urinary incontinence.

Outcome measures:

The primary objective of the study is to evaluate the effect of tolterodine 4 mg on the nocturnal incontinence. This will be done by comparing the effect of the drug in the same group and by comparing its effect between different groups.

Sample size:

Assuming type I statistical error of 5 % and type II statistical error of 20 %, we designed our study to have a power of 80 %. Based on the results of the previous studies, the expected difference between the study and control group is 59- 70 %.15, 17The dropped out number of cases is suspected to be 10-20%. So, the sample size required to give significant difference is 60 in each arm.

Statistical analysis:

The ICIQ- UI score, number of pads and the number of nocturnal incontinence episodes will be expressed as mean± SD. Independent sample T-test will be used for comparison of means. All statistical tests will be done using Statistical Package for the Social Sciences 16.0 for Microsoft (SPSS, Inc., Chicago, Illinois, USA) with a p value of less than 0.05 considered significant.

The protocol is accepted by the local ethical committee of Faculty of medicine, Mansoura University ( Mansoura Faculty of Medicine- Institutional Research Board MFM-IRB) and given the number of R/16.07.51 Figure 1: study design and time schedule

ELIGIBILITY:
Inclusion Criteria:

* Patients who passed at least one year follow up after the procedure.
* Patients who have no symptoms or signs of oncological failure (local recurrence or distant metastasis).
* Presence of NI with normal daytime continence assessed by the Arabic version of short form International Consultation on Incontinence questionnaire (ICIQ-UI Short Form).18
* Normal renal function (eGFR ˃50 ml/min /1.73m2) calculated by the Modification Of Diet in Renal Disease study equation.
* Ability to provide informed consent.

Exclusion Criteria:

* Patients who did not pass one year postoperative.
* Presence of oncological failure.
* Totally continent patient or who has daytime incontinence or chronic urine retention.
* Impaired renal function.
* Uncontrolled DM or hypertension.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-05; Primary Completion 2017-11 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
improvement of nocturnal incontinence | 10 weeks
  the score of ICIQ- UI short form questionnaire

REFERENCES:
- [Derived] Zahran MH, Harraz AM, Taha DE, Nabeeh H, El Hefnawy AS, Ali-El-Dein B. The short-term effects of tolterodine on nocturnal incontinence after ileal orthotopic neobladder: a randomised crossover placebo-controlled study. BJU Int. 2019 Oct;124(4):679-686. doi: 10.1111/bju.14769. Epub 2019 Apr 22. PMID 30946525